CLINICAL TRIAL: NCT07137104
Title: A Phase I/IIa Study to Investigate the Safety, Tolerability, and Preliminary Effectiveness of HeXell-2020 in Patients With Stable Coronary Artery Disease (CAD)
Brief Title: Safety and Preliminary Effectiveness Study of Mesenchymal Stem Cells, HeXell-2020, in Patients With Stable Coronary Artery Disease
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hexun Biosciences Co., LTD. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HEXUMBA20221222
Record Dates: First submitted 2025-07-17; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-07

CONDITIONS: Coronary Artery Disease
Keywords: HeXell-2020; Coronary Artery Disease (CAD); Mesenchymal Stem Cells (MSC)
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: Phase I: Single arm, 2 dose cohorts with dose-defining escalation Phase IIa: Single arm, with dose determined in Phase I
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment Cohort (Experimental): Phase 1 ：single arm. two cohort. cohort 1: HeXell-2020 will be administered by intravenous once every two weeks, and a total of 3 doses.
  cohort 2: HeXell-2020 will be administered by intravenous once every two weeks, and a total of 6 doses.
  Phase 2a: Single arm.
  Interventions: Drug: HeXell-2020

INTERVENTIONS:
Drug: HeXell-2020 — Phase I Cohort 1: HeXell-2020 with a total of 3 doses, 9x10^7 cells/dose.
  Phase I Cohort 2: HeXell-2020 with a total of 6 doses, 9x10^7 cells/dose.
  Phase IIa: RP2D from phase I.

SUMMARY:
This is a phase I/IIa study to investigate the safety, tolerability, and preliminary effectiveness of HeXell-2020 in patients with stable coronary artery disease (CAD). HeXell-2020 is an investigational drug product consisting of allogenic umbilical cord mesenchymal stem cells (UCMSCs) as the drug substance. All enrolled and eligible subjects will receive HeXell-2020 treatment.

DETAILED DESCRIPTION:
Coronary artery disease (CAD) is the most common form of heart disease and a leading cause of mortality worldwide. It is a manifestation of myocardial ischemia, a condition resulting from insufficient blood flow to the myocardial tissue. CAD occurs when the coronary arteries become progressively narrowed and stiffened due to atherosclerosis-the accumulation of cholesterol, lipids, and plaque along the inner arterial walls. Narrowed blood vessels and increased shear stress may contribute to plaque destabilization, vessel outward remodeling, as well as increased pro-inflammatory cytokines production, leading to advanced atherosclerosis. As the disease advances, this narrowing impairs coronary blood flow, causing permanent heart damage. Over time, CAD can progressively weaken the heart muscle, contributing to heart failure.

Mesenchymal stem cells (MSC) become a potential therapeutic tool for treating cardiovascular diseases due to their capabilities in tissue repair, anti-oxidation, immune-modulation and anti-inflammatory. Intravenous infusion of HeXell-2020, the allogenic umbilical cord MSC, in an atherosclerotic rat model improved blood glucose tolerance, LDL cholesterol levels, and the severity of aortic arch stenosis. Additionally, results further demonstrated significant improvement in atherosclerotic lesions caused by fat deposition at the aortic arch and descending aorta after the treatment. Although the mode of actions of MSCs in CADs have not been fully elucidated, these nonclinical results, together with the established immunomodulatory and anti-inflammatory effects of MSCs, are supportive for the rationale of HeXell-2020 in treating patients with CAD.

This study is composed of two phases, Phase I and Phase IIa. In Phase I, two cohorts were designed following traditional 3+3 scheme to define recommended phae 2 dose (RP2D). In Phase IIa, 22 evaluable subjects are estimated. Safety and efficacy will be evaluated through follow-up visit over one year.

ELIGIBILITY:
Inclusion Criteria:

1. Subject who is able to understand the nature of this study and accepts to enter the study by signing written informed consent
2. Male or female who are aged between 18 and 75 years old on date of consent
3. Patient without LV thrombus or ventricular aneurysm documented by echocardiography at screening
4. Patient having a diagnosis of CAD caused by ≥ 50% stenosis of at least 1 major or larger epicardial coronary artery (target vessel ≥ 2 mm in diameter without in-stent restenosis) documented by imaging studies within 12 months prior to the date of dosing. If the stenosis results are derived from CCTA, the examination time of CCTA should be at least 6 months prior to screening.
5. Patient with Canadian Cardiovascular Society (CCS) Class I, II, or III angina pectoris and received optimal, stable, medical therapy (e.g., anticoagulants therapy, β-blockers, calcium channel blockers, nitrates, ranolazine) per country specific treatment guidelines for at least 4 weeks prior to the date of screening, if prescribed
6. Patients with stable hemodynamic parameters and adequate pulmonary function, defined as systolic pressure ≥ 90 mmHg and < 150 mmHg, and heart rate > 50/min and <110/min on at least 2 consecutive readings, at screening and baseline (before dosing)
7. Patient's medical history shows no history of organ or cell transplant rejection, or suspected contraindication to HeXell-2020 including the components (penicillin and streptomycin).
8. Female subjects show negative pregnancy test results within 30 days prior to the first study treatment.
9. All male patients and female patients with child-bearing potential (between puberty and 2 years after menopause) should use at least any one of the appropriate contraception methods shown below, during dosing and for at least 4 weeks after stopping study treatment.

   1. Total abstinence (when this is in line with the preferred and usual lifestyle of the subject). Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.
   2. Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy), total hysterectomy, or tubal ligation at least 6 weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment.
   3. Male sterilization (at least 6 months prior to screening). For female subjects on the study, the vasectomized male partner should be the sole partner for that subject.
   4. Combination of any two of the following listed methods: (d.1+d.2 or d.1+d.3, or d.2+d.3):

   d.1. Use of oral, injected or implanted hormonal methods of contraception or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception. Please refer to 8.2 Prohibited Treatments for detailed information.

   d.2. Placement of an intrauterine device (IUD) or intrauterine system (IUS). d.3. Barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical/vault caps).

Exclusion Criteria:

1. Subject had participated in investigational drug trials and took any investigational drugs within 28 days prior to the first treatment.
2. Patient is schedule to [or has received within 180 days prior to Screening Visit] undergo the following coronary revascularization throughout the study period:

   * Coronary artery bypass grafting (CABG)
   * Valve repair/replacement
   * Cardiac resynchronization therapy (CRT) device
3. Patient is scheduled to undergo percutaneous coronary intervention (PCI) during the trial before screening.
4. Patient with high-risk or unstable acute coronary syndrome (e.g., myocardial infarction), major cardiovascular surgery (e.g., coronary valve replacement, or aortic aneurysm surgery), stroke, transient ischemic attack (TIA), carotid surgery, pulmonary embolism, or deep venous thrombosis in past 90 days prior to the date of screening
5. Patient with evidence of medical condition as follows,

   * Acute cardiac decompensation
   * Congenital heart disease
   * Significantly uncorrected valvular heart disease
   * Malignant arrhythmia in the absence of a defibrillator
   * Severe pulmonary disease
   * Essential thrombocytosis
   * Anti-phospholipid syndrome
   * Other hypercoagulable disorders (e.g., disseminated intravascular coagulation, Factor V Leiden)
6. Patient with poorly controlled diabetes mellitus (HbA1c >8%) or a known history or present evidence of conditions that may affect study assessments (e.g., currently receiving chemotherapeutic or immunosuppressant agents, or have received prior radiation therapy to the chest)
7. Patient carry history of malignancy of any organ system (other than curatively treated localized basal or squamous cell carcinoma of the skin, cervical carcinoma in situ, or superficial bladder cancer) within 5 years prior to study entry.
8. Subject had a history of drug abuse or alcohol abuse according to the Diagnostic and Statistical Manual of Mental Disorders 5th edition (DSM-5) criteria.
9. Evidence of inadequate hematopoietic, hepatic, and renal function as determined by any one of the following laboratory requirements:

   * Hemoglobin <8.5 mg/dL
   * Estimated glomerular filtration rate (eGFR) <45 mL/min/1.73 m2 as calculated by the Modified in Diet in Renal Disease (MDRD) formula or requiring dialysis prior to study dosing.
   * Total bilirubin >2× upper limit of normal (ULN)
   * Alanine aminotransferase (ALT) >3× ULN
10. Patient with HIV, active HBV, or active HCV infections
11. Subject who is pregnant or lactating
12. Subject with underlying medical, mental or psychological conditions that would impair the treatment compliance, unable to undergo study-required tests/scans for any reason, or in the opinion of the investigator would not permit to participate in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of TEAE, SAE and SUSAR over the study | Within the first year after cell transplantaion
  To evaluate the number of treatment emergent adverse events (TEAEs), serious adverse events (SAEs), suspected and unexpected serious adverse reactions (SUSARs) over the study period,
To determine the recommended phase II dose (RP2D) in Phase I study | Within the first year after cell transplantaion
  To determination RP2D, number and proportion of subjects having experienced DLTs will be presented and the RP2D should be determined on the indicated dose at which ≤ 1 patient experiences DLT out of 6 patients who have been DLT evaluated.
Change in myocardial perfusion defect severity under the rest acquisition and pharmacological stress of dipyridamole in Phase IIa study | Before first dosing and at 12 months post cell transplantaion
  Measured by SPECT with thallium-201 from baseline. The SRS, SSS and SDS are three variables used to measure cardiac perfusion and ischemia.

SECONDARY OUTCOMES:
Time to the first occurrence of major adverse cardiovascular events (MACEs) | From the date of the first treatment until the first occurrence of MACE, death, or study cut-off point, unless the subject has withdrawn consent for all contacts or is loss of follow-up, whichever came first, assessed up to 24 months.
  Including AMI, stroke, cardiovascular mortality, and hospitalization for unstable angina or revascularization procedures, from the date of the first treatment will be analyzed by Kaplan-Meier method.
Change in the evaluation result of CCTA from baseline | Before first dosing and at 3, 6 months post cell transplantation
  The stenosis percent of the different coronary segments, using the 17-segment model.
Change from baseline in echocardiographic measures. | Before first dosing and at 3, 6, 12 months post cell transplantation
  Ventricular remodeling: including LVEF in percentage, global longitudinal strain (GLS) in percentage.
Change in functional class of angina by using CCS angina classification from baseline. | Before first dosing, and 1, 3, 6 , 12 months post cell transplantation
  Change in functional class of angina by using CCS angina classification will be summarized descriptively by visit
Change in the 6-minute walk test (6-MWT) from baseline. | Before first dosing and 6, 12 months post cell transplantation
  The 6-MWT measures the distance walked on level ground in 6 minutes.
Change in serum levels of amino-terminal pro-brain natriuretic peptide (NT pro-BNP) and high sensitivity cardiac troponin (hs-cTn) from baseline. | Before first dosing, and 1, 3, 6 , 12 months post cell transplantation
  Change in serum levels of NT pro-BNP and hs-cTn from baseline will be summarized descriptively.
Change in quality of life using the Seattle Angina Questionnaire (SAQ) from baseline. | Before first dosing, and 1, 3, 6 , 12 months post cell transplantation
  The SAQ, a 19-item self-administered questionnaire measuring 5 dimensions of CAD: physical limitation, anginal stability, anginal frequency, treatment satisfaction and disease perception will be used to assess the functional change of CAD in HeXell-2020 administered patients.
Change from baseline in echocardiographic measures. | Before first dosing and at 3, 6, 12 months post cell transplantation
  Myocardial performance [including isovolumic relaxation time (IVRT), isovolumic contraction time (IVCT), LV ejection time (ET), and myocardial performance index (MPI or Tei Index)][MPI= (IVCT+IVRT)/ET]
Change in the evaluation result of CCTA from baseline | Before first dosing and at 3, 6 months post cell transplantation
  Severity of stenosis assessed by 2022 Coronary Artery Disease Reporting and Data System (CAD-RADSTM 2.0), ranging from CAD-RADS 0 for absence of any plaque or stenosis to CAD-RADS 5 for the presence of at least 1 totally occluded coronary artery.
Change in the evaluation result of CCTA from baseline | Before first dosing and at 3, 6 months post cell transplantation
  Coronary artery calcium score (CACS, as per Agatston method, J Am Coll Cardiol. 1990;15:827-32), higher scores mean a worse outcome.
Change from baseline in echocardiographic measures. | Before first dosing and at 3, 6, 12 months post cell transplantation.
  Ventricular remodeling: LV end-diastolic volume (EDV) in mL, and end-systolic volume (ESV) in mL, stroke volume (SV in ), calculated by EDV - ESV ( mL)
Change from baseline in echocardiographic measures. | Before first dosing and at 3, 6, 12 months post cell transplantation.
  Ventricular remodeling: LV internal diameter in diastole and systole (LVIDd and LVIDs in mm), interventricular septum diameter (IVSD in mm), posterior wall thickness (PWT in mm), anteroseptal wall thickness (ASWT in mm)

IPD SHARING:
Plan to Share IPD: No